CLINICAL TRIAL: NCT01826474
Title: A Phase IIb, Open-label Study to Assess the Efficacy, Safety, Pharmacodynamics and Pharmacokinetics of Multiple Subcutaneous Doses of PRO045 in Subjects With Duchenne Muscular Dystrophy
Brief Title: Phase IIb Study of PRO045 in Subjects With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO045-CLIN-01
Record Dates: First submitted 2013-03-20; First posted 2013-04-08 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; DMD; Prosensa; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- PRO045, cohort 1 (Experimental): 0.15 mg/kg until dose-titration
  Interventions: Drug: PRO045, 0.15 mg/kg/week
- PRO045, cohort 2 (Experimental): 1.0 mg/kg until dose-titration
  Interventions: Drug: PRO045, 1.0 mg/kg/week
- PRO045, cohort 3 (Experimental): 3.0 mg/kg until dose-titration
  Interventions: Drug: PRO045, 3.0 mg/kg/week
- PRO045, cohort 4 (Experimental): 6.0 mg/kg until dose-titration
  Interventions: Drug: PRO045, 6.0 mg/kg/week
- PRO045, cohort 5 (Experimental): 9.0 mg/kg until move to 48 week treatment phase
  Interventions: Drug: PRO045, 9.0 mg/kg/week
- PRO045, cohort 6 (Experimental): 48 week treatment phase
  Interventions: Drug: PRO045, selected dose

INTERVENTIONS:
Drug: PRO045, 0.15 mg/kg/week — Subcutaneous injection
  Arms: PRO045, cohort 1
Drug: PRO045, 1.0 mg/kg/week — Subcutaneous injection
  Arms: PRO045, cohort 2
Drug: PRO045, 3.0 mg/kg/week — Subcutaneous injection
  Arms: PRO045, cohort 3
Drug: PRO045, 6.0 mg/kg/week — Subcutaneous injection
  Arms: PRO045, cohort 4
Drug: PRO045, 9.0 mg/kg/week — Subcutaneous injection
  Arms: PRO045, cohort 5
Drug: PRO045, selected dose — Subcutaneous injection
  Arms: PRO045, cohort 6

SUMMARY:
The purpose of the study is to see whether PRO045 is safe and effective to use as medication for Duchenne Muscular Dystrophy (DMD) patients with a mutation around location 45 in the DNA for the dystrophin protein.

DETAILED DESCRIPTION:
A phase IIb, open-label, multiple-dose study. The study consists of two phases; a dose escalation phase (with subsequent dose-titration) and a 48-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Duchenne muscular dystrophy resulting from a mutation correctable by treatment with PRO045 confirmed by a state-of-the-art DNA diagnostic technique covering all DMD gene exons, including but not limited to MLPA (Multiplex Ligation-dependent Probe Amplification), CGH (Comparative Genomic Hybridisation), SCAIP (Single Condition Amplification/Internal Primer) or HRMCA (High-Resolution Melting Curve Analysis), and correctable by PRO045-induced DMD exon 45 skipping in cultured skin-derived myo-converted fibroblasts.
2. Ambulant boys aged at least 5 years on the day of first dosing able to walk for at least 230 meters in the 6 minute walking distance (6MWD) test at first screening visit and also at the baseline visit. In addition, 2 of the 3 pre-treatment 6MWD tests (screen 1, screen 2, baseline) must be within +/-30 metres of each other prior to first PRO045 administration.
3. Adequate quality for biopsy (confirmed with MRI) of the lateral head of the gastrocnemius muscle. An alternative muscle may be considered for biopsy but only following discussion between the Principal Investigator and the Prosensa Medical Monitor.
4. Life expectancy of at least 3 years after inclusion in the study.
5. Glucocorticosteroid use which is stable for at least 3 months prior to first PRO045 administration. Subjects must have been receiving glucocorticosteroids for at least 6 months prior to the first PRO045 administration.
6. Willing and able to adhere to the study visit schedule and other protocol requirements.
7. Written informed consent signed (by parent(s)/legal guardian and/or the subject, according to the local regulations).
8. In France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

1. Known presence of dystrophin in ≥5% of fibres in a pre-study diagnostic muscle biopsy (i.e. historic muscle biopsy taken prior to written informed consent for this study).
2. Current or history of liver disease or impairment.
3. Current or history of renal disease or impairment.
4. At least two aPTT above ULN within the last month.
5. Screening platelet count below the lower limit of normal (LLN).
6. Acute illness within 4 weeks prior to first dose of PRO045 which may interfere with the study assessments.
7. Severe mental retardation or behavioural problems which in the opinion of the investigator prohibits participation in this study.
8. Severe cardiomyopathy which in the opinion of the investigator prohibits participation in this study. If a subject has a left ventricular ejection fraction <45% at screening, the investigator should discuss inclusion of the subject with the Medical Monitor.
9. Expected need for daytime mechanical ventilation within the next year.
10. Use of anticoagulants, antithrombotics or antiplatelet agents.
11. Use of idebenone or other forms of coenzyme Q10 within 1 month prior to the start of the screening for the study.
12. Use of nutritional or herbal supplements which, in the opinion of the investigator, may influence muscle performance, within 1 month of the study.
13. Use of any other investigational product or participation in another trial with an investigational product, within 6 months prior to the start of the screening for the study.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 6 minute walk test | after 48 weeks of treatment phase

SECONDARY OUTCOMES:
Muscle function | after 48 weeks of treatment phase
Muscle strength | after 48 weeks treatment phase
Performance of upper limb | after 48 weeks of treatment phase
Functional outcomes questionnaire | after 48 weeks of treatment
Safety | after 48 weeks of treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: T. Voit, MD PhD, Principal Investigator — Institut de Myologie
Locations (6):
- UZ Leuven, Leuven, Belgium
- Institut de Myologie, Paris, France
- Policlinico Universitario Agostino Gemelli, Roma, Italy
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - Institute of Genetic Medicine International Centre for Life, Newcastle

REFERENCES:
- See also: BioMarin website — http://www.biomarin.com